CLINICAL TRIAL: NCT06415136
Title: Adjacent Level Anterior Cervical Fusion: SeaSpine Shoreline Versus Removal of Previously Implanted Plate and Replating
Status: Enrolling by invitation | Type: Observational
Sponsor: Research Source (Network)
Responsible Party: Sponsor
Other Study IDs: SeaSpine-001
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Degenerative Disc Disease; Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Degeneration; Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- SeaSpine Shoreline: All enrolled patients will receive the SeaSpine Shoreline device.
  Interventions: Device: SeaSpine Shoreline

INTERVENTIONS:
Device: SeaSpine Shoreline — The SeaSpine Shoreline device is a minimally invasive cervical plate/cage system.

SUMMARY:
The purpose of this study is to evaluate the efficacy of SeaSpine Shoreline device in surgery of the cervical spine.

DETAILED DESCRIPTION:
This is a retrospective, prospective, post-market, observational, single-center, single surgeon study evaluating the use of the SeaSpine Shoreline device. Patients will be identified by the Investigator as needing, or already received the device during a cervical fusion surgery and meeting all the inclusion and none of the exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Appropriate patient, as determined by the Investigator, scheduled for an elective cervical spine fusion to treat adjacent level cervical disc herniation or degeneration resulting in cervical radiculopathy or myelopathy
2. At least 18 years of age
3. Failure of nonoperative care
4. Previous anterior cervical plating
5. Psychosocially, mentally and physically able to comply with this protocol including adhering to follow-up schedule and study requirements

Exclusion Criteria:

1. Pregnancy or anticipated to become pregnant during the course of the study
2. No previous cervical spine surgery
3. Non-instrumented cervical fusion
4. Cervical fusion with separate plate fixation
5. Unwilling or unable to sign consent
6. Patient has any condition, that in the opinion of the Investigator, would prohibit the patient from complying with the protocol
7. Currently a prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A patient who meets all inclusion criteria and none exclusion criteria will be enrolled in the study. A patient is considered enrolled upon placement of the SeaSpine Shoreline device during the surgical procedure. If the surgeon decides intra-operatively not to utilize the SeaSpine Shoreline device, the patient will be considered a screen failure.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Cervical fusion assessed via CT scan | 12 months post surgery
  Motion, bridging on radiograph, and bridging bone on CT scan
Clinical outcome via neck visual analog scale (VAS) | 12 months post surgery
  Standard of care patient reported neck visual analog scale (VAS) will be used to evaluate patient pain. On a scale of 0 to 10 with a score of 0 being no pain and a score of 10 being worst pain. A low score means a better clinical outcome. A high score means a worse clinical outcome.
Clinical outcome via neck disability index (NDI) | 12 months post surgery
  Standard of care patient reported neck disability index (NDI) will be used to evaluate patient pain and quality of life. On a vertical scale of 0 to 5 with a score of 0 meaning neck pain (if any) does not interfere with life activities and 5 meaning neck pain strongly interferes with life activities. A low score means a better clinical outcome. A high score means a worse clinical outcome.
Clinical outcome via Dysphagia score | 12 months post surgery
  Standard of care patient reported dysphagia score will be used to evaluate patient inability or difficulty swallowing. On a scale of 0 to 4 with a score of 0 meaning no difficulty and 4 meaning severe problem. A low score means a better clinical outcome. A high score means a worse clinical outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Michigan Orthopaedic Surgeons, Southfield, Michigan, United States